CLINICAL TRIAL: NCT06143527
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for the Treatment of Polycystic Ovary Syndrome
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for PCOS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023MSC-01
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Polycystic Ovary Syndrome; PCOS
Keywords: Polycystic Ovary Syndrome (PCOS); Polycystic Ovary Syndrome; PCOS; Stem Cell; Stem Cells; Mesenchymal Stem Cells; Umbilical Cord Derived Mesenchymal Stem Cells
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): Intravenous infusion
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — Cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of cultured allogeneic adult umbilical cord derived mesenchymal stem cells delivered intravenously for the treatment of Polycystic Ovary Syndrome.

DETAILED DESCRIPTION:
Stem cell treatment has shown efficacy for PCOS in both human and animal studies. Complete resolution was seen of polycystic ovary syndrome (PCOS) in a young woman after a single intravenous injection of umbilical cord derived mesenchymal stem cells (UCDSC). It is hypothesized that intravenous infusion of UCDSC can reduce or eliminate PCOS. Patients will receive roughly 2 million umbilical cord derived mesenchymal stem cells per kg of body weight. Hormone levels and ultrasound will be checked 3,6 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

• Ultrasound documented poly cystic ovary syndrome

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety
* Continued drug abuse
* Previous organ transplant
* Hypersensitivity to sulfur
* Inability to supply proper informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2027-11-16 (Estimated); Study Completion 2027-11-16 (Estimated)

PRIMARY OUTCOMES:
Safety: Adverse Events | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: Global Improvement Score (GI) | Four year follow-up
  Ranging from 0 to 100%

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick C Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Athens Beverly Hills Medical Group, Glyfada, Greece

IPD SHARING:
Plan to Share IPD: No